CLINICAL TRIAL: NCT07107373
Title: MavAcamten Real World eVidEnce coLlaboration in HCM (MARVEL-HCM)
Brief Title: A Study to Assess the Treatment of Obstructive Hypertrophic Cardiomyopathy (oHCM) With Mavacamten in the US
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV027-1152
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy (oHCM)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants receiving treatment mavacamten
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Mavacamten — According to the product label

SUMMARY:
The purpose of this study is to evaluate the real-world safety and effectiveness of patients with symptomatic obstructive hypertrophic cardiomyopathy (oHCM) initiated on mavacamten at certain high volume HCM centers in the US

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the index date
* Prescription of mavacamten for the treatment of Obstructive hypertrophic cardiomyopathy (oHCM) with NYHA Class II or III
* ≥ 12 weeks of follow-up after prescription of mavacamten, except for the baseline data reporting

Exclusion Criteria:

* Data collection as part of a clinical trial during the study period
* Participation in a myosin inhibitor clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise of adult individuals diagnosed with Obstructive hypertrophic cardiomyopathy (oHCM) that have been prescribed mavacamten treatment between April 29th, 2022, and August 6th, 2024
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
New York Heart Association (NYHA) functional class | Baseline, and at weeks 4, 8, 12, 24, 36, 48, 60, 72, and in increments of 12 weeks thereafter from index
Left ventricular outflow tract (LVOT) gradient and associated parameters | Baseline, and at weeks 4, 8, 12, 24, 36, 48, 60, 72, and in increments of 12 weeks thereafter from index
Left ventricular ejection fraction (LVEF) and associated parameters | Baseline, and at weeks 4, 8, 12, 24, 36, 48, 60, 72, and in increments of 12 weeks thereafter from index

SECONDARY OUTCOMES:
Mavacamten dose at initiation | Day 1
Mavacamten dose change | Up to 72 weeks
Reason for mavacamten dose change | Up to 72 weeks
Reason for mavacamten permanent discontinuation | Up to 72 weeks
Reason for treatment interruption | Up to 72 weeks
Prior Obstructive hypertrophic cardiomyopathy (oHCM) therapies | Baseline
Concurrent Obstructive hypertrophic cardiomyopathy (oHCM) therapies | Up to 72 weeks
Other cardiovascular-related treatments prescribed | Up to 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- University of California, San Francisco (UCSF), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts